CLINICAL TRIAL: NCT02269332
Title: Association of 25-OH Vitamin D Status With Findings on Screening Colonoscopy.
Brief Title: Vitamin D and Screening Colonoscopy or Polyp Surveillance
Acronym: VitDColon
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20140085H
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening Colonoscopy: Referred for a screening colonoscopy or polyp surveillance or had one in the last 2 weeks
  Interventions: Other: Screening Colonoscopy

INTERVENTIONS:
Other: Screening Colonoscopy — we will obtain serum vitamin D blood levels from those scheduled for a screening colonoscopy or polyp surveillance

SUMMARY:
The investigators will recruit DoD beneficiaries 18 years or older, that have been referred for a screening colonoscopy or polyp surveillance (or had one in the last 2 weeks), and have no previous diagnosis of colorectal cancer. They will have a 25 OH Vitamin D level drawn to determine if there is an association between the level obtained and findings on colonoscopy, or previous findings (if repeating).

DETAILED DESCRIPTION:
DoD beneficiaries age 18 or older will be recruited from the clinics at the Mike O'Callaghan Federal Medical Center (MOFMC). Subjects meeting the inclusion/exclusion criteria will be offered an opportunity to participate:

Screening Visit:

* Obtain signed Informed Consent Document and HIPAA Authorization (research-driven).
* Record: Date of birth, age, gender, race, ethnicity, current email address, height (in inches), weight (in pounds), waist circumference (in inches) measurement, blood pressure, and whether subject is taking or has taken any vitamin D supplement or derivative, and if so, note the dosage, frequency, and duration of therapy.
* Subjects will be told to fast for at least 10 hours prior to Visit 1

Visit 1 (within two weeks of their screening colonoscopy):

-Subjects will have the following research-driven blood test drawn which include: Serum 25-OH vitamin D via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood will be drawn)

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* DoD beneficiaries 18 years or older
* Referred for a screening colonoscopy or polyp surveillance or had one in the last 2 weeks

Exclusion:

* Previous diagnosis of colorectal cancer, adenomatous polyps, and/or cancer
* Military trainees
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DoD beneficiaries age 18 or older will be recruited from the clinics at the Mike O'Callaghan Federal Medical Center (MOFMC). Subjects meeting the inclusion/exclusion criteria will be offered an opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Bryce, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Hospital/Nellis Air Force Base, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Screening Colonoscopy
Started | 298
Completed | 228 (number analyzed)
Not Completed | 70

BASELINE CHARACTERISTICS:
Arm/Group | Screening Colonoscopy
Number analyzed (Participants) | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 298
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 164

OUTCOME MEASURES:

1. Primary Outcome: Serum Vitamin D
Description: Vitamin D blood levels will be obtained at the time of procedure.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Colonoscopy
Number analyzed (Participants) | 228
Participants
  vitamin D insufficiency (<30ng/ml) | 155
  vitamin D normal (>30ng/ml) | 73

2. Primary Outcome: Adenomatous Polyps
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Colonoscopy
Number analyzed (Participants) | 228
Participants
  found to have adenomatous polyps | 104
  did not have adenomatous polyps | 124

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Screening Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/298
Serious Adverse Events (participants affected / at risk) | 0/298
Other Adverse Events (participants affected / at risk) | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes